CLINICAL TRIAL: NCT01073033
Title: Oral Supplement for Pregnant and Lactating Mothers to Promote Infant Immune Maturation and Protection Against Early Life Infections
Brief Title: Oral Supplement for Pregnant and Lactating Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08.10 INF
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Diarrhea; Acute Respiratory Infection
Keywords: pregnancy; lactation; oral supplement; probiotics; early infections
MeSH Terms: conditions — Diarrhea; Breast Feeding; Infections | interventions — Gravidity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- oral supplement1 (Experimental): Oral supplement for pregnant and lactating mothers
  Interventions: Dietary Supplement: milk supplement 1
- oral supplement 2 (Active Comparator): Oral supplement for pregnant and lactating mothers
  Interventions: Dietary Supplement: milk supplement 2
- Reference (No Intervention): No oral supplementation during pregnancy and lactating.

INTERVENTIONS:
Dietary Supplement: milk supplement 1 — milk supplement with probiotics
  Other Names: Suitable for pregnant and lactating period.
  Arms: oral supplement1
Dietary Supplement: milk supplement 2 — milk supplement without probiotics
  Other Names: Suitable for pregnant and lactating periode.
  Arms: oral supplement 2

SUMMARY:
To assess protection against early life infections through supplementation of mothers during pregnancy to the newborns' growth, morbidity, immune status intra and extra-uterine.

DETAILED DESCRIPTION:
During pregnancy mothers have to fulfill the tremendous physiological needs to support their own immune status as well as that of their babies. Accordingly, it appears highly valuable to provide mothers with a nutritional supplement during pregnancy and lactation to promote the immune development in newborns, thus reinforcing the infants' defenses.

In that respect, an appropriate maternal diet must provide sufficient energy and nutrients to meet the mother's usual requirements and promote health status, as well as the needs of the growing fetus and beyond for the neonate.

Key organogenesis steps take place during fetal life and many functional features of the immune system are already coded in the genetic asset of the individual. However, at birth the immune system remains fairly immature. An epigenetic, postnatal instruction seems to be extremely important for the maturation of the immune system allowing its full functionality.

The cross-talk between the mother and her baby is, indeed, crucial for the optimal development of the foetus and subsequently for the full and functional maturation of the neonate.

The newborn relies for his protection almost exclusively on his innate immune system that is initially instructed and educated early in life by factors derived from his mother as well as post-natal environmental factors such as early life colonization with micro-organisms that activates the innate immunity and enhance Th1-cell polarization thereby potentially reducing atopic dermatitis with respect to the hygiene hypothesis.

A large part of this immune education is provided by factors transmitted from the mother pre-natally through the placenta or post-natally via the breast milk. Breast milk contains a number of nutrients and bioactive components, including immune cells, maternal antibodies (mainly secretory IgA), cytokines, growth factors, lactoferrin, nucleotides, triacylglycerols, fatty acids, oligosaccharides, and vitamins. All together, these components beneficially impact the health status of the newborn, conferring, among other functions, immune education and early protection.

A typical example of such transfer of immune competence is the TGF-β that could be transmitted in active from either through the placenta or absorbed by the neonates through the milk. This TGF-β is an important IgA switch factor and this is likely to be responsible, in part, for the capacity of breast-fed infant to produce higher levels of mucosal SIgA compared to non-breast fed infants. Moreover, milk soluble CD14 transmitted to the newborn contributes to prime the neonatal gut to modulate the microbial recognition and establishment of endogenous microbiota.

Diarrhea episodes are major manifestation of common infant infections of viral or bacterial aetiology and are a key health concern in paediatrics. As mentioned above there are evidences that some probiotic strains significantly improve diarrheal outcomes in infants, particularly rotavirus diarrhea. In that respect diarrhea occurrence was selected as the primary outcome in the present trial.

ELIGIBILITY:
Inclusion Criteria:

* Expecting mothers who are in their 6th month of pregnancy
* Willing to consume 2 x 200 ml of test product daily
* Willing to exclusively breastfeed until the baby is at least 2-month old
* Having signed the informed consent

Exclusion Criteria:

* Known allergy to cow's milk
* Subjects previously diagnosed HIV(+) and Hepatitis B (+)
* Multiple pregnancy
* High risk pregnancy (pre-eclampsia, diabetes, etc)
* Currently participating or having participated in another clinical trial during the last 3 months
* Subjects who consumed pro- and /or prebiotics-containing food/supplement* in the month before inclusion

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The incidence of diarrhea in infants from birth to 1 year | 24 months

SECONDARY OUTCOMES:
In infants: growth, morbidity, immune maturation, metabolomics profile | 18 months
In mothers: fetal growth, general health, immune system, metabolomics profile and preterm delivery | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Valerie Guinto, MD, Principal Investigator — University of the Philippines; Dr. Jacinto Mantaring, MD, Principal Investigator — University of the Philippines
Locations (1):
- Ospital Ng Muntinlupa, Manila, Philippines

REFERENCES:
- [Derived] Mantaring J, Benyacoub J, Destura R, Pecquet S, Vidal K, Volger S, Guinto V. Effect of maternal supplement beverage with and without probiotics during pregnancy and lactation on maternal and infant health: a randomized controlled trial in the Philippines. BMC Pregnancy Childbirth. 2018 May 31;18(1):193. doi: 10.1186/s12884-018-1828-8. PMID 29855271